CLINICAL TRIAL: NCT04749771
Title: A Scaleable Video Coaching Intervention for Opioid-using Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 256792
Record Dates: First submitted 2021-02-01; First posted 2021-02-11 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Child Behavior; Parent-Child Relations; Substance Use; Substance Abuse
Keywords: parent training; early adversity; early intervention; manualized intervention; high-risk children; parenting; fMRI
MeSH Terms: conditions — Child Behavior; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two groups. Half of the participants will be randomized into the experimental condition (FIND) while the other half will be randomized into the active control condition (HTP)
Who Masked: Participant
Masking Description: Research assistants collecting the data during lab visits will not know the condition of the participant and will therefore not be biased during data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filming Interactions to Nurture Development (FIND) (Experimental): FIND is a brief video coaching intervention which involves feedback provided by the coach to the caregiver using brief film clips derived from video of caregiver-child interaction. The coaching focuses on showing caregivers instances in which they are engaging in developmentally-supportive interactions during coaching sessions. FIND is delivered over 10 weekly sessions lasting 30-45 minutes. The process begins with an initial session in which the coach provides an overview, records 10-15 minutes of caregiver-child interaction, then introduces the concept of serve and return. The video is edited to show brief clips in which the caregiver is engaged in the first of five specific caregiver-based components of serve and return. The next week, the FIND coach reviews the edited clips in detail with the caregiver. Sessions continue, alternating between filming and coaching sessions until all five components have been covered sequentially.
  Interventions: Behavioral: Filming Interactions to Nurture Development
- The Healthy Toddler Program (HTP) (Active Comparator): HTP, the active control intervention, consists of weekly sessions alternating between (a) coaching sessions covering one of five domains of child development (Motor, Cognitive, Language, Play, and Social-Emotional and (b) observation sessions that will include a review of the prior coaching session and an observation and discussion of the caregiver-child interaction. This intervention will consist of 10 sessions each lasting 25-30 minutes. The coach will not engage in any filming or video coaching, but will be able to discuss caregiving concerns. HTP materials are adapted from the Partners for a Healthy Baby curriculum developed by Florida State University's Center for Prevention and Early Intervention Policy.
  Interventions: Behavioral: The Healthy Toddler Program

INTERVENTIONS:
Behavioral: Filming Interactions to Nurture Development — FIND is a brief video coaching intervention which involves feedback provided by the coach to the caregiver using brief film clips derived from video of caregiver-child interaction collected in the home.
  Other Names: FIND
  Arms: Filming Interactions to Nurture Development (FIND)
Behavioral: The Healthy Toddler Program — HTP, the active control intervention, consists of weekly sessions alternating between (a) coaching sessions covering one of five domains of child development (Motor, Cognitive, Language, Play, and Social-Emotional and (b) observation sessions that will include a review of the prior coaching session and an observation and discussion of the caregiver-child interaction.
  Other Names: HTP
  Arms: The Healthy Toddler Program (HTP)

SUMMARY:
This study will adapt and evaluate a novel, innovative, and highly scalable parenting intervention that employs video coaching to target responsive parenting, Filming Interactions to Nurture Development (FIND), among women who have been referred to or are in treatment for opioid misuse/addiction.

DETAILED DESCRIPTION:
The overall objective of this study is to conduct a randomized trial with a sample of opioid-using women who are in or have been referred for treatment through outpatient and inpatient services and have a child aged 0-36 months. We will use a longitudinal design with an active control condition to test the central hypothesis that associations between (a) increases in responsive caregiving and (b) subsequent caregiver opioid addiction recovery, psychological well-being, and child developmental and biobehavioral outcomes (secondary targets), will be partially mediated through (c) changes in caregiver executive functioning, reward responsiveness, and parent self-concept. The rationale for this work is that it simultaneously addresses the unmet needs of a large, significantly underserved population and allows for a rigorous test of our conceptual model, which specifies hypothesized underlying mechanisms and differential impact.

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult (18-50 years of age)
* Must be the biological parent of a child between the ages of 0-48 months of age
* Must have received, or be currently receiving, treatment for a substance use disorder for any DSM-5 class of substance use disorder except caffeine or tobacco. This includes alcohol, cannabis, hallucinogens, inhalants, opioids, sedatives, hypnotics/anxiolytics, and stimulants.
* Must have their child at least two days each week at study entry

Exclusion Criteria:

* Metal implants, metal fragments, pacemakers, or other electronic medical implants
* Claustrophobic
* Weigh > 550 lbs
* Women who are or think they may be pregnant
* History of neurological disorders
* Left-handed

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of parenting stress via the Parent Stress Index-IV | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  Items are on a 5-point scale ranging from "strongly agree" to "strongly disagree." Higher scores indicated greater parenting stress.
  The measures includes three subscales and a total score:
  * Parental distress (12 items) sum score ranging between 12-60
  * Parent-child dysfunctional interaction (12 items) sum score ranging between 12-60
  * Difficult child (12 items) sum score ranging between 12-60
  * Total score (36 items) sum score ranging between 36-180
Caregiver's perceived sense of competency in parenting via the Parent Sense of Competency scale (PSOC) | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The Parenting Sense of Competence (PSOC) questionnaire is filled out by the caregiver to assess parents' sense of competence and enjoyment of parenting. This is an adapted version of the PSOC (original PSOC has 17 items, Johnston & Mash, 1989), with 18 items and simplified language for lower reading levels.
  These items are answered on a 4-point scale ranging from "strongly agree" to "strongly disagree." Scoring for some items is reversed so that, for all items, higher scores indicate greater parenting self-esteem. Nine (9) items (#s 2,3,4,5,8,9,13,15 and 17) on the PSOC are reverse coded.
  Subscales include:
  Satisfaction: Mean score of 2,3,4,5,9,13,15,17, and 18 (Range = 1-4) Efficacy: Mean score of 1,6,7,8,10,11,14, and 16 (Range = 1-4) Total Score: 18 - 72, scored responses summed
Assessment of the caregivers motivation via measurement on the Behavioral Inhibition System and Behavioral Activation System (BIS/BAS) scale | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The BIS/BAS Scale is a 24-item self-report questionnaire designed to measure two motivational systems: the behavioral inhibition system (BIS) and the behavioral activation system (BAS). Participants respond to each item using a 4-point Likert scale. The scale has four subscales.
  One subscale corresponds to the BIS. Seven items contribute to this score. The remaining three subscales correspond to three components of BAS.
  BAS Drive measures the motivation to follow one's goals. Four items contribute to this score.
  BAS Reward Responsiveness measures the sensitivity to pleasant reinforcers in the environment. Four items contribute to this score.
Assessment of emotional or behavioral problems in children as assessed by the SDQ-Infant questionnaire | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire. 25 items are asked on a 3-point scale from not-true to certainly true. Followed by 5 items assessing difficulties with emotions, concentration, behavior or being able to get along with people.
Measurement of Opioid Craving via Opioid Craving Scale | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The Opioid Craving Scale is a modification of the Cocaine Craving Scale (Weiss et al., 1995, 1997, 2003) used to measure opioid craving. The scale consists of three items rated on a visual analogue scale from 0-10
Self-report of income, occupation and financial strain via the ECHO measure (Income, Occupation, Financial Strain) | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  This measure is a 9-item self-report of income, occupation and financial strain.
Measurement of social support via the Social Support Questionnaire | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  Measures social support, yielding scores for:
  * Perceived number of social supports
  * Satisfaction with social support that is available Questionnaire consists of 27 items with 2-part responses (listing the people they can turn to and rely upon and how satisfied they are with the social supports).
  Each item is scored based on the number of support persons listed, and the satisfaction scale scored on a scale of 1 to 6 (1 = very satisfied and 6 = very dissatisfied). The overall number and satisfaction scores are summed and divided by 27.
Self-report of commitment and support in regards to family members as assessed by the Cohesion subscale of the Family Enviornment Scale | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The Family Environment Scale (FES) is a self-report 90-item instrument developed to assess the social climates of families focusing on the measurement and description of interpersonal relationships among family members on the directions of personal growth and the basic organizational structure of the family.
  The Cohesion subscale is a 9-item scale intended to measue the degree of commitment and support that family members provide each other. Respondents rate statements on a scale from mostly true to mostly false.
Communicative skills assessed via the MacArthur Communicative Development Inventories (MCDI) | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The MacArthur Communicative Development Inventories (MCDI) are parent- report instruments for assessing communicative skills in infants and toddlers.
  The infant form (Level I), designed for children between 8 and 18 months, contains an 89-word vocabulary checklist with separate columns for comprehension and production. There are two equivalent forms of the toddler form (Level II, Forms A and B), both designed for children between 16 and 30 months. Each form contains 100 vocabulary items.
  Use appropriate norming tables for girls and boys to furnish raw score values for every 5th percentile level from the 5th to the 99th rank.
Observed level of inhibitory control via the Stop Signal Task | Change from baseline at endpoint (3-4 months post-baseline)
  Inhibitory control will be assessed by the Stop Signal Task (SST) during an MRI scan. The task speed adjusts based on performance and a single response time score will be outputted for each participant. The key neural measure is the degree of blood oxygenation-level dependent (BOLD) signal during stop trials relative to go trials (i.e., the "stop > go" contrast over the entire trial period).
Observed Parental Self-Concept | Change from baseline at endpoint (3-4 months post-baseline)
  The PSET involves visual presentation of single words or short phrases in the parenting domain (e.g., kind, supportive, enforces rules) seen under two different instruction conditions. The identity condition will ask participants to indicate via a button press whether the word or phrase describes them as a parent (left index finger = yes, right index finger = no). The control condition will ask participants to indicate via a button press whether the word or phrase is a quality that can change for a parent (yes/no). Scores are percent endorsement of developmentally-supportive (DS) and developmentally-unsupportive (DU) items in each condition. The key neural contrasts are neural activation during the presentation of (a) identity > control trials and (b) identity-yes > identity-no trials.
Coded rate of responsive caregiving via conversational turns | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  Conversational turns is a simple coding scheme designed to record timing, quantity, and length of caregiver and child utterances.
Assessment of parent's warmth and hostility towards their child through the use of the Iowa Family Interaction Rating Scales | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  The Iowa family interaction rating scales were used to assess parent's warmth and hostility towards their partner, their perceived warmth and hostility received from their partner, and warmth and hostility towards their child. The questionnaire is divided into 3 parts; the first 10 questions ask how you have behaved towards your partner, the next 10 ask how your partner has behaved towards you, and the final 10 questions ask how you have behaved towards your child.
  There are 2 scales for each part of the questionnaire, warmth (6 items) and hostility (4 items). For both scales each item has a possible 7 responses. Each scale reverse scored and then summed by adding each item score, giving a possible range of 0-42 for the warmth scale and 0-28 for the hostility scale. Higher scores indicate higher levels of warmth/hostility respectively.

SECONDARY OUTCOMES:
Mobile Messaging for Responsive Caregiving (MMRC) | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  Caregiver's self-reported rate of responsive caregiving interactions between child and caregiver.
Demographic information | Baseline
  Demographic information including socioeconomic status, age and sex of caregiver and child, education level, race/ethnicity
Incidence of early adversity assessed via the Adverse Childhood Experiences (ACEs) | Baseline
  The ACE is a 10-item measure of childhood adversity and is often used as a predicter of poorer outcomes later in life. The higher the score out of 10, the more likely for poor outcomes.
  Sum the scores of all responses 1-10 for total ACE score. Reverse code the emotional neglect question, question 10, which counts as an ACE if either sub-question is answered "No." The developers suggest not including the supplemental questions in the Total ACE score. They recommend remaining true to the original ACE 10 categories so we can compare data across sites. If desired, you can sum the scores on the supplementary questions, and create a supplementary grand total to examine separately.
  TotalACES=total ACE score TotalSupp=sum of supplemental questions TotalAll=Sum of ACE score and supplemental question score
Assessment of mental health domains across psychiatric conditions via the use of the PhenX Broad Psychopathology questionnaire | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  This measure consists of 23 questions that assess 13 psychiatric domains, including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. Each item inquires about how much (or how often) the individual has been bothered by the specific symptom during the past 2 weeks.
Intervention Fidelity assessed through use of a fidelity criteria rubric | Assessed at the conclusion of the intervention, directly before endpoint (3-4 months post-baseline)
  Intervention Fidelity is assessed by the number of required items completed from a checklist of required actions for the given intervention.
Intervention Dosage as assessed by number of sessions complete | Assessed at the conclusion of the intervention, directly before endpoint (3-4 months post-baseline)
  Intervention Dosage is assessed by the number of completed sessions for each intervention.
  Total FIND Sessions Complete = Count of sessions complete (0-10) Total HTP Sessions Complete = Count of sessions complete (0-10)
Assessment of unpredictability and fragmentation of early-life environments in infants and children through the use of the Questionnaire of Unpredictability in Childhood (QUIC) | At Baseline
  The QUIC, a reliable and valid self-report assessment of exposure to unpredictability in the social, emotional, and physical domains during early life, is a brief, comprehensive, and promising instrument for predicting risk for mental illness. The QUIC consists of an overall score and five separate subscale scores. Higher scores indicate more exposure to unpredictability in childhood. To obtain the overall score or subscale scores, reverse score select items (indicated by an R after the item number) and then calculate the sum of the items in each scale: Parental monitoring and involvement = 1R + 3R + 4R + 5R + 6R + 7R + 9R + 10R + 14R Parental predictability = 2 + 8R + 11 + 12 + 15R + 16 + 17R + 31 + 32 + 33 + 34 + 35 Parental environment = 18 + 19 + 21 + 22 + 28R + 29 + 30 Physical environment = 13 + 20 + 26 + 27 + 36R + 37 + 38 Safety and security = 23 + 24 + 25 Overall = Sum of all subscales.
Self-reported substance use and treatment history as assessed by questionnaire modified from PhenX and iOpen | Change from baseline at endpoint (3-4 months post-baseline) and 6 months post-endpoint
  Questionnaire developed from PhenX and iOpen to assess substance use and treatment history.

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Fisher, Ph.D., Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data collected from the study will be eligible for sharing externally. Audio/Video cannot be shared due to confidentiality, however data coded from these types of files will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Eligible IPD will be made available 1-year after the study is complete.
Access Criteria: IPD access requests must be approved by the study's Principal Investigator, Dr. Philip Fisher. Requests should include information about who will be given access to the IPD and what the IPD will be used for. If approved, a Data Use Agreement (DUA) will need to be completed between the University of Oregon and the institution where the IPD will be sent.

REFERENCES:
- [Background] National Institutes of Health. Improve Treatments for Opioid Misuse and Addiction: NIH Heal Intitiative. 2018; https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/improve-treatments-opioid-misuse-addiction. Accessed September 17, 2018.
- [Background] Patrick SW, Davis MM, Lehmann CU, Cooper WO. Increasing incidence and geographic distribution of neonatal abstinence syndrome: United States 2009 to 2012. J Perinatol. 2015 Aug;35(8):650-5. doi: 10.1038/jp.2015.36. Epub 2015 Apr 30. PMID 25927272
- [Background] National Institutes of Health. HEAL Initiative Research Plan. 2018; https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/heal-initiative-research-plan. Accessed September 17, 2018.
- [Background] National Institute on Drug Abuse. Dramatic Increases in Maternal Opioid Use and Neonatal Abstinence Syndrome. 2015; https://www.drugabuse.gov/related-topics/trends-statistics/infographics/dramatic-increases-in-maternal-opioid-use-neonatal-abstinence-syndrome. Accessed September 17, 2018.
- [Background] Patrick SW, Schumacher RE, Benneyworth BD, Krans EE, McAllister JM, Davis MM. Neonatal abstinence syndrome and associated health care expenditures: United States, 2000-2009. JAMA. 2012 May 9;307(18):1934-40. doi: 10.1001/jama.2012.3951. Epub 2012 Apr 30. PMID 22546608
- [Background] Rutherford HJV, Barry DT, Mayes LC. Family-Focused Approaches to Opioid Addiction Improve the Effectiveness of Treatment. 2018; https://www.srcd.org/policy-media/child-evidence-briefs/opioid-addiction. Accessed September 18, 2018.
- [Background] Luby JL. Poverty's Most Insidious Damage: The Developing Brain. JAMA Pediatr. 2015 Sep;169(9):810-1. doi: 10.1001/jamapediatrics.2015.1682. No abstract available. PMID 26191940
- [Background] Maheu FS, Dozier M, Guyer AE, Mandell D, Peloso E, Poeth K, Jenness J, Lau JY, Ackerman JP, Pine DS, Ernst M. A preliminary study of medial temporal lobe function in youths with a history of caregiver deprivation and emotional neglect. Cogn Affect Behav Neurosci. 2010 Mar;10(1):34-49. doi: 10.3758/CABN.10.1.34. PMID 20233954
- [Background] Shaw DS, Vondra JI. Infant attachment security and maternal predictors of early behavior problems: a longitudinal study of low-income families. J Abnorm Child Psychol. 1995 Jun;23(3):335-57. doi: 10.1007/BF01447561. PMID 7642841
- [Background] Quevedo K, Waters TE, Scott H, Roisman GI, Shaw DS, Forbes EE. Brain activity and infant attachment history in young men during loss and reward processing. Dev Psychopathol. 2017 May;29(2):465-476. doi: 10.1017/S0954579417000116. PMID 28401835
- [Background] Blair C, Raver CC. Poverty, Stress, and Brain Development: New Directions for Prevention and Intervention. Acad Pediatr. 2016 Apr;16(3 Suppl):S30-6. doi: 10.1016/j.acap.2016.01.010. PMID 27044699
- [Background] Wachs TD, Georgieff M, Cusick S, McEwen BS. Issues in the timing of integrated early interventions: contributions from nutrition, neuroscience, and psychological research. Ann N Y Acad Sci. 2014 Jan;1308:89-106. doi: 10.1111/nyas.12314. Epub 2013 Dec 19. PMID 24354763
- [Background] Lowell DI, Carter AS, Godoy L, Paulicin B, Briggs-Gowan MJ. A randomized controlled trial of Child FIRST: a comprehensive home-based intervention translating research into early childhood practice. Child Dev. 2011 Jan-Feb;82(1):193-208. doi: 10.1111/j.1467-8624.2010.01550.x. PMID 21291437
- [Background] Gardner F, Shaw DS, Dishion TJ, Burton J, Supplee L. Randomized prevention trial for early conduct problems: effects on proactive parenting and links to toddler disruptive behavior. J Fam Psychol. 2007 Sep;21(3):398-406. doi: 10.1037/0893-3200.21.3.398. PMID 17874925
- [Background] Shaw DS, Dishion TJ, Supplee L, Gardner F, Arnds K. Randomized trial of a family-centered approach to the prevention of early conduct problems: 2-year effects of the family check-up in early childhood. J Consult Clin Psychol. 2006 Feb;74(1):1-9. doi: 10.1037/0022-006X.74.1.1. PMID 16551138
- [Background] Shonkoff JP, Fisher PA. Rethinking evidence-based practice and two-generation programs to create the future of early childhood policy. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1635-53. doi: 10.1017/S0954579413000813. PMID 24342860
- [Background] Rutherford HJV, Potenza MN, Mayes LC. The neurobiology of addiction and attachment. In: Suchman N, Pajulo M, Mayes LC, eds. Parents and Substance Addiction: Developmental Approaches to Intervention. New York, NY: Oxford University Press; 2013.
- [Background] Rutherford HJ, Williams SK, Moy S, Mayes LC, Johns JM. Disruption of maternal parenting circuitry by addictive process: rewiring of reward and stress systems. Front Psychiatry. 2011 Jul 6;2:37. doi: 10.3389/fpsyt.2011.00037. eCollection 2011. PMID 21779252
- [Background] Patterson G. Coercive Family Process. Eugene, OR: Castalia Publishing Company; 1982.
- [Background] Patterson GR, Reid JB. Social interactional processes within the family: The study of the moment-by-moment family transactions in which human social development is imbedded. J Appl Dev Psychol. 1984;5(3):237-262.
- [Background] Buggey T, Ogle L. Video self-modeling. Psychol Schs. 2012;49(1):52-70.
- [Background] Dowrick PW. A review of self modeling and related interventions. Appl Prev Psychol. 1999;8(1):23-39.
- [Background] Fisher PA, Burraston B, Pears K. The early intervention foster care program: permanent placement outcomes from a randomized trial. Child Maltreat. 2005 Feb;10(1):61-71. doi: 10.1177/1077559504271561. PMID 15611327
- [Background] Sweller J. Cognitive Load During Problem Solving: Effects on Learning. Cogn Sci. 1988;12(2):257-285
- [Background] Sweller J, Van Merrienboer JJG, Paas FGWC. Cognitive architecture and instructional design. Educ Psychol Rev. 1998;10(3):251-296.
- [Background] Mayer RE, Moreno R. Nine Ways to Reduce Cognitive Load in Multimedia Learning. Educ Psychol. 2003;38(1):43-52
- [Background] Bryck RL, Fisher PA. Training the brain: practical applications of neural plasticity from the intersection of cognitive neuroscience, developmental psychology, and prevention science. Am Psychol. 2012 Feb-Mar;67(2):87-100. doi: 10.1037/a0024657. Epub 2011 Jul 25. PMID 21787037
- [Background] Shonkoff JP, Garner AS; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. The lifelong effects of early childhood adversity and toxic stress. Pediatrics. 2012 Jan;129(1):e232-46. doi: 10.1542/peds.2011-2663. Epub 2011 Dec 26. PMID 22201156
- [Background] Shonkoff JP, Bales SN. Science does not speak for itself: translating child development research for the public and its policymakers. Child Dev. 2011 Jan-Feb;82(1):17-32. doi: 10.1111/j.1467-8624.2010.01538.x. PMID 21291426
- [Background] Fisher PA, Gunnar MR, Dozier M, Bruce J, Pears KC. Effects of therapeutic interventions for foster children on behavioral problems, caregiver attachment, and stress regulatory neural systems. Ann N Y Acad Sci. 2006 Dec;1094:215-25. doi: 10.1196/annals.1376.023. PMID 17347353
- [Background] Dozier M, Albus K, Fisher PA, Sepulveda S. Interventions for foster parents: implications for developmental theory. Dev Psychopathol. 2002 Fall;14(4):843-60. doi: 10.1017/s0954579402004091. PMID 12549706
- [Background] Flannery JE, Beauchamp KG, Fisher PA. The role of social buffering on chronic disruptions in quality of care: evidence from caregiver-based interventions in foster children. Soc Neurosci. 2017 Feb;12(1):86-91. doi: 10.1080/17470919.2016.1170725. Epub 2016 Apr 19. PMID 27021231
- [Background] Hser YI, Hoffman V, Grella CE, Anglin MD. A 33-year follow-up of narcotics addicts. Arch Gen Psychiatry. 2001 May;58(5):503-8. doi: 10.1001/archpsyc.58.5.503. PMID 11343531
- [Background] Martin-Soelch C, Chevalley AF, Kunig G, Missimer J, Magyar S, Mino A, Schultz W, Leenders KL. Changes in reward-induced brain activation in opiate addicts. Eur J Neurosci. 2001 Oct;14(8):1360-8. doi: 10.1046/j.0953-816x.2001.01753.x. PMID 11703464
- [Background] Fisher PA, Chamberlain P. Multidimensional treatment foster care: A program for intensive parenting, family support, and skill building. J Emot Behav Disord. 2000;8(3):155-164.
- [Background] Leve LD, Harold GT, Chamberlain P, Landsverk JA, Fisher PA, Vostanis P. Practitioner review: Children in foster care--vulnerabilities and evidence-based interventions that promote resilience processes. J Child Psychol Psychiatry. 2012 Dec;53(12):1197-211. doi: 10.1111/j.1469-7610.2012.02594.x. Epub 2012 Aug 6. PMID 22882015
- [Background] Thomas R, Zimmer-Gembeck MJ. Behavioral outcomes of Parent-Child Interaction Therapy and Triple P-Positive Parenting Program: a review and meta-analysis. J Abnorm Child Psychol. 2007 Jun;35(3):475-95. doi: 10.1007/s10802-007-9104-9. Epub 2007 Feb 27. PMID 17333363
- [Background] Sanders MR, Kirby JN, Tellegen CL, Day JJ. The Triple P-Positive Parenting Program: a systematic review and meta-analysis of a multi-level system of parenting support. Clin Psychol Rev. 2014 Jun;34(4):337-57. doi: 10.1016/j.cpr.2014.04.003. Epub 2014 Apr 26. PMID 24842549
- [Background] Furlong M, McGilloway S, Bywater T, Hutchings J, Smith SM, Donnelly M. Behavioural and cognitive-behavioural group-based parenting programmes for early-onset conduct problems in children aged 3 to 12 years. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD008225. doi: 10.1002/14651858.CD008225.pub2. PMID 22336837
- [Background] Suchman NE, DeCoste C, Castiglioni N, McMahon TJ, Rounsaville B, Mayes L. The Mothers and Toddlers Program, an attachment-based parenting intervention for substance using women: post-treatment results from a randomized clinical pilot. Attach Hum Dev. 2010 Sep;12(5):483-504. doi: 10.1080/14616734.2010.501983. PMID 20730641
- [Background] Suchman NE, DeCoste CL, McMahon TJ, Dalton R, Mayes LC, Borelli J. Mothering From the Inside Out: Results of a second randomized clinical trial testing a mentalization-based intervention for mothers in addiction treatment. Dev Psychopathol. 2017 May;29(2):617-636. doi: 10.1017/S0954579417000220. PMID 28401850
- [Background] Fukkink RG. Video feedback in widescreen: a meta-analysis of family programs. Clin Psychol Rev. 2008 Jul;28(6):904-16. doi: 10.1016/j.cpr.2008.01.003. Epub 2008 Feb 5. PMID 18359136
- [Background] Balldin S, Fisher PA, Wirtberg I. Video feedback intervention with children: A systematic review. Res Soc Work Pract. 2016:1049731516671809.
- [Background] O'Hara L, Smith ER, Barlow J, Livingstone N, Herath NI, Wei Y, Spreckelsen TF, Macdonald G. Video feedback for parental sensitivity and attachment security in children under five years. Cochrane Database Syst Rev. 2019 Nov 29;11(11):CD012348. doi: 10.1002/14651858.CD012348.pub2. PMID 31782528
- [Background] Bakermans-Kranenburg MJ, van IJzendoorn MH, Juffer F. Less is more: meta-analyses of sensitivity and attachment interventions in early childhood. Psychol Bull. 2003 Mar;129(2):195-215. doi: 10.1037/0033-2909.129.2.195. PMID 12696839
- [Background] Schindler HS, Fisher PA, Shonkoff JP. From Innovation to Impact at Scale: Lessons Learned From a Cluster of Research-Community Partnerships. Child Dev. 2017 Sep;88(5):1435-1446. doi: 10.1111/cdev.12904. Epub 2017 Aug 4. PMID 28777436
- [Background] Lippard CN, Riley KL, Hughes-Belding K. OBSERVING TODDLERS' INDIVIDUAL EXPERIENCES IN CLASSROOMS: INITIAL USE OF THE PARENTING INTERACTIONS WITH CHILDREN: CHECKLIST OF OBSERVATIONS LINKED TO OUTCOMES. Infant Ment Health J. 2016 Sep;37(5):549-59. doi: 10.1002/imhj.21584. Epub 2016 Aug 24. PMID 27554914
- [Background] Abidin RR. Parenting Stress Index-Short Form. Pediatric Psychology Press Charlottesville, VA; 1990.
- [Background] Johnston C, Mash EJ. A measure of parenting satisfaction and efficacy. J Clin Child Psychol. 1989;18(2):167-175.
- [Background] Bethell C, Gombojav N, Solloway M, Wissow L. Adverse Childhood Experiences, Resilience and Mindfulness-Based Approaches: Common Denominator Issues for Children with Emotional, Mental, or Behavioral Problems. Child Adolesc Psychiatr Clin N Am. 2016 Apr;25(2):139-56. doi: 10.1016/j.chc.2015.12.001. Epub 2016 Jan 11. PMID 26980120
- [Background] Carroll JE, Gruenewald TL, Taylor SE, Janicki-Deverts D, Matthews KA, Seeman TE. Childhood abuse, parental warmth, and adult multisystem biological risk in the Coronary Artery Risk Development in Young Adults study. Proc Natl Acad Sci U S A. 2013 Oct 15;110(42):17149-53. doi: 10.1073/pnas.1315458110. Epub 2013 Sep 23. PMID 24062432
- [Background] Smith KE, Landry SH, Swank PR. The influence of decreased parental resources on the efficacy of a responsive parenting intervention. J Consult Clin Psychol. 2005 Aug;73(4):711-20. doi: 10.1037/0022-006X.73.4.711. PMID 16173858
- [Background] Theise R, Huang KY, Kamboukos D, Doctoroff GL, Dawson-McClure S, Palamar JJ, Brotman LM. Moderators of intervention effects on parenting practices in a randomized controlled trial in early childhood. J Clin Child Adolesc Psychol. 2014;43(3):501-9. doi: 10.1080/15374416.2013.833095. Epub 2013 Sep 24. PMID 24063291
- [Background] Brophy-Herb HE, Gibbons C, Omar MA, Schiffman RF. Low-income fathers and their infants: Interactions during teaching episodes. Infant Ment Health J. 1999;20(3):305-321.
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Chamberlain P, Reid JB. Parent observation and report of child symptoms. Behav Assess. 1987.
- [Background] Zimmerman IL, Steiner VG, Pond RE. PLS-5: Preschool Language Scales. Bloomington, MN: Pearson/Psychological Corporation; 2012.
- [Background] Barlow J, Johnston I, Kendrick D, Polnay L, Stewart-Brown S. Individual and group-based parenting programmes for the treatment of physical child abuse and neglect. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD005463. doi: 10.1002/14651858.CD005463.pub2. PMID 16856097
- [Background] Fisher PA, Skowron EA. Social-learning parenting intervention research in the era of translational neuroscience. Curr Opin Psychol. 2017 Jun;15:168-173. doi: 10.1016/j.copsyc.2017.02.017. Epub 2017 Mar 16. PMID 28813257
- [Background] Piquero AR, Farrington DP, Welsh BC, Tremblay R, Jennings WG. Effects of early family/parenting programs on antisocial behavior and. Campbell Syst Rev. 2008;11.
- [Background] McDermott JM, Pears KC, Bruce J, Kim HK, Roos L, Yoerger KL, Fisher PA. Improving kindergarten readiness in children with developmental disabilities: Changes in neural correlates of response monitoring. Appl Neuropsychol Child. 2018 Jul-Sep;7(3):187-199. doi: 10.1080/21622965.2017.1286239. Epub 2017 Feb 22. PMID 28631968
- [Background] Bruce J, McDermott JM, Fisher PA, Fox NA. Using behavioral and electrophysiological measures to assess the effects of a preventive intervention: a preliminary study with preschool-aged foster children. Prev Sci. 2009 Jun;10(2):129-40. doi: 10.1007/s11121-008-0115-8. PMID 19030992
- [Background] Giuliani NR, Beauchamp KG, Fisher PA. Inhibitory control mechanisms of a nurturing parenting intervention. Society for Research on Child Development April 6-8, 2017; Austin, TX.
- [Background] Verbruggen F, Logan GD. Response inhibition in the stop-signal paradigm. Trends Cogn Sci. 2008 Nov;12(11):418-24. doi: 10.1016/j.tics.2008.07.005. PMID 18799345
- [Background] Noll LK, Giuliani NR, Beauchamp KG, Fisher PA. Behavioral and neural correlates of parenting self-evaluation in mothers of young children. Soc Cogn Affect Neurosci. 2018 May 1;13(5):535-545. doi: 10.1093/scan/nsy031. PMID 29718429
- [Background] Diekhof EK, Falkai P, Gruber O. Functional neuroimaging of reward processing and decision-making: a review of aberrant motivational and affective processing in addiction and mood disorders. Brain Res Rev. 2008 Nov;59(1):164-84. doi: 10.1016/j.brainresrev.2008.07.004. Epub 2008 Jul 21. PMID 18675846
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631
- [Background] Luijten M, Schellekens AF, Kuhn S, Machielse MW, Sescousse G. Disruption of Reward Processing in Addiction : An Image-Based Meta-analysis of Functional Magnetic Resonance Imaging Studies. JAMA Psychiatry. 2017 Apr 1;74(4):387-398. doi: 10.1001/jamapsychiatry.2016.3084. PMID 28146248
- [Background] Gross TJ, Mason WA, Parra G, Oats R, Ringle J, Haggerty KP. Adherence and Dosage Contributions to Parenting Program Quality. J Soc Social Work Res. 2015 Dec;6(4):467-489. doi: 10.1086/684108. PMID 26726301
- [Background] Axford N, Bywater T, Blower S, Berry V, Baker V, Morpeth L. Critical factors in the successful implementation of evidence-based parenting programmes: Fidelity, adaptation and promoting quality. In L. Dixon, d.F. Perkins, C. Hamilton-Giachritsis, L.A. Craig, eds.: The Wiley Handbook of What Works in Child Maltreatment: An Evidence-Based Approach to Assessment and Intervention in Child Protection. Hoboken, NJ: Wiley-Blackwell; 2017:349-366.
- [Background] Walker CK, Tancredi DJ, Bennett D, Halladay A, Butler R, Schmidt RJ. The Early Life Exposures Assessment Tool (ELEAT). Unpublished instrument. Davis, CA: University of California, Davis; 2013.
- [Background] Chandler P, Sweller J. Cognitive load theory and the format of instruction. Cogn Instruct. 1991;8(4):293-332.
- [Background] Mayer RE, Heiser J, Lonn S. Cognitive constraints on multimedia learning: When presenting more material results in less understanding. J Educ Psychol. 2001;93(1):187-198. doi: 110.1037/0022-0663.1093.1031.1187.
- [Background] Mousavi SY, Low R, Sweller J. Reducing cognitive load by mixing auditory and visual presentation modes. J Educ Psychol. 1995;87(2):319.
- [Background] Baddeley A. Working memory: theories, models, and controversies. Annu Rev Psychol. 2012;63:1-29. doi: 10.1146/annurev-psych-120710-100422. Epub 2011 Sep 27. PMID 21961947
- [Background] Baddeley AD. Working memory. Phil Trans R Soc Lond B. 1983;302(1110):311-324.
- [Background] Smith EE, Jonides J. Storage and executive processes in the frontal lobes. Science. 1999 Mar 12;283(5408):1657-61. doi: 10.1126/science.283.5408.1657. PMID 10073923
- [Background] Kellam, S. G., & Rebok, G. W. (1992). Building developmental and etiological theory through epidemiologically based preventive intervention trials. In J. McCord & R. E. Tremblay (Eds.), Preventing Antisocial Behavior: Interventions From Birth Through Adolescence (pp. 162-195). New York, NY, US: Guilford Press.
- [Background] Fisher PA. Translational Neuroscience as a Tool for Intervention Development in the Context of High-Adversity Families. New Dir Child Adolesc Dev. 2016 Sep;2016(153):111-25. doi: 10.1002/cad.20165. PMID 27589501
- [Background] Fisher PA, Frenkel TI, Noll LK, Berry M, Yockelson M. Promoting Healthy Child Development via a Two-Generation Translational Neuroscience Framework: The Filming Interactions to Nurture Development Video Coaching Program. Child Dev Perspect. 2016 Dec;10(4):251-256. doi: 10.1111/cdep.12195. Epub 2016 Aug 10. PMID 28936231
- [Background] Love JM, Kisker EE, Ross C, Raikes H, Constantine J, Boller K, Brooks-Gunn J, Chazan-Cohen R, Tarullo LB, Brady-Smith C, Fuligni AS, Schochet PZ, Paulsell D, Vogel C. The effectiveness of early head start for 3-year-old children and their parents: lessons for policy and programs. Dev Psychol. 2005 Nov;41(6):885-901. doi: 10.1037/0012-1649.41.6.88. PMID 16351335
- [Background] Roggman LA, Cook GA, Innocenti MS, Jump Norman V, Christiansen K. Parenting interactions with children: Checklist of observations linked to outcomes (PICCOLO) in diverse ethnic groups. Infant Ment Health J. 2013;34(4):290-306.
- [Background] Melby JN, Conger RD. The Iowa family interaction rating scales: Instrument summary. In: Kerig PK, Lindahl KM, eds. Family Observational Coding Systems. New York, NY: Psychology Press; 2000:49-74.
- [Background] RTI International. PhenX Toolkit. 24.0 ed. www.phenxtoolkit.org: RTI International; 2018.
- [Background] Flannery BA, Volpicelli JR, Pettinati HM. Psychometric properties of the Penn Alcohol Craving Scale. Alcohol Clin Exp Res. 1999 Aug;23(8):1289-95. PMID 10470970
- [Background] Rosenberg H. Clinical and laboratory assessment of the subjective experience of drug craving. Clin Psychol Rev. 2009 Aug;29(6):519-34. doi: 10.1016/j.cpr.2009.06.002. Epub 2009 Jun 11. PMID 19577831
- [Background] Narrow WE, Clarke DE, Kuramoto SJ, Kraemer HC, Kupfer DJ, Greiner L, Regier DA. DSM-5 field trials in the United States and Canada, Part III: development and reliability testing of a cross-cutting symptom assessment for DSM-5. Am J Psychiatry. 2013 Jan;170(1):71-82. doi: 10.1176/appi.ajp.2012.12071000. PMID 23111499
- [Background] Baron IS. Behavior rating inventory of executive function. Child Neuropsychol. 2000 Sep;6(3):235-8. doi: 10.1076/chin.6.3.235.3152. No abstract available. PMID 11419452
- [Background] Carver CS, White TL. Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: the BIS/BAS scales. J Personality Soc Psychol. 1994;67(2):319.
- [Background] Torrubia R, Avila C, Moltó J, Caseras X. The Sensitivity to Punishment and Sensitivity to Reward Questionnaire (SPSRQ) as a measure of Gray's anxiety and impulsivity dimensions. J Personality Indiv Diff. 2001;31(6):837-862.
- [Background] Gartstein MA, Rothbart MK. Studying infant temperament via the revised infant behavior questionnaire. J Infant Behav Dev. 2003;26(1):64-86.
- [Background] Putnam SP, Gartstein MA, Rothbart MK. Measurement of fine-grained aspects of toddler temperament: the early childhood behavior questionnaire. Infant Behav Dev. 2006 Jul;29(3):386-401. doi: 10.1016/j.infbeh.2006.01.004. Epub 2006 Mar 2. PMID 17138293
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Briggs-Gowan M, Carter A. Brief Infant-Toddler Social and Emotional Assessment (BITSEA) manual, version 2.0. New Haven, CT: Yale University; 2002.
- [Background] Hane AA, LaCoursiere JN, Mitsuyama M, Wieman S, Ludwig RJ, Kwon KY, V Browne J, Austin J, M Myers M, Welch MG. The Welch Emotional Connection Screen: validation of a brief mother-infant relational health screen. Acta Paediatr. 2019 Apr;108(4):615-625. doi: 10.1111/apa.14483. Epub 2018 Aug 13. PMID 29959878
- [Background] Fan J, McCandliss BD, Fossella J, Flombaum JI, Posner MI. The activation of attentional networks. Neuroimage. 2005 Jun;26(2):471-9. doi: 10.1016/j.neuroimage.2005.02.004. Epub 2005 Mar 19. PMID 15907304
- [Background] Eriksen BA, Eriksen CW. Effects of noise letters upon the identification of a target letter in a nonsearch task. Percept Psychophys. 1974;16(1):143-149.
- [Background] van Veen V, Cohen JD, Botvinick MM, Stenger VA, Carter CS. Anterior cingulate cortex, conflict monitoring, and levels of processing. Neuroimage. 2001 Dec;14(6):1302-8. doi: 10.1006/nimg.2001.0923. PMID 11707086
- [Background] Jankowski KF, Moore WE, Merchant JS, Kahn LE, Pfeifer JH. But do you think I'm cool? Developmental differences in striatal recruitment during direct and reflected social self-evaluations. Dev Cogn Neurosci. 2014 Apr;8:40-54. doi: 10.1016/j.dcn.2014.01.003. Epub 2014 Jan 26. PMID 24582805
- [Background] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899
- [Background] Smith CT, Wallace DL, Dang LC, Aarts E, Jagust WJ, D'Esposito M, Boettiger CA. Modulation of impulsivity and reward sensitivity in intertemporal choice by striatal and midbrain dopamine synthesis in healthy adults. J Neurophysiol. 2016 Mar;115(3):1146-56. doi: 10.1152/jn.00261.2015. Epub 2015 Dec 16. PMID 26683066
- [Background] Bell RP, Yi JY, Chen Y, et al. Activity based reward processing among opiate users: Validation of the behavioral incentive delay task. J Drug Alcohol Depend. 2017;171:e17-e18.
- [Background] Winter C, Dishion TJ. Parent Consultant Log. Eugene, OR: Prevention Science Institute; 2007.
- [Background] Fisher P, Greenley K, Pears K. Service Utilization Interview. Unpublished measure. In:1999.
- [Background] Moos R, Moos B. Family Environment Scale Manual: Development, Applications, Research. Third ed. Palo Alto, CA: Consulting Psychologist Pres; 1994.
- [Background] Teicher MH, Parigger A. The 'Maltreatment and Abuse Chronology of Exposure' (MACE) scale for the retrospective assessment of abuse and neglect during development. PLoS One. 2015 Feb 25;10(2):e0117423. doi: 10.1371/journal.pone.0117423. eCollection 2015. PMID 25714856
- [Background] Sterne JA, White IR, Carlin JB, Spratt M, Royston P, Kenward MG, Wood AM, Carpenter JR. Multiple imputation for missing data in epidemiological and clinical research: potential and pitfalls. BMJ. 2009 Jun 29;338:b2393. doi: 10.1136/bmj.b2393. PMID 19564179
- [Background] Berkman ET, Reise SP. A Conceptual Guide to Statistics Using SPSS. Sage; 2011.